CLINICAL TRIAL: NCT06959745
Title: Magnesium-L-Threonate Improves Menopausal Symptoms: A Single-center, Single-blind, Randomized, Placebo-Controlled Pilot Study
Brief Title: Magnesium-L-Threonate Improves Menopausal Symptoms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Jie Li, Professor, Deputy director of global health research center, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2025-240-02
Record Dates: First submitted 2025-04-25; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Menopause Syndrome; Magnesium
Keywords: menopause syndrome
MeSH Terms: interventions — threonic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium-L-Threonate (Experimental)
  Interventions: Drug: Magnesium-L-Threonate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Magnesium-L-Threonate — Magnesium L-threonate, 1740 mg, taken orally, twice a day, for 8 weeks.
  Arms: Magnesium-L-Threonate
Drug: Placebo — Placebo, 1740 mg, taken orally, twice a day, for 8 weeks.
  Arms: Placebo

SUMMARY:
This trial has a randomized, single-blind, single-center, parallel-controlled design, with participant screening and trial implementation conducted at Guangdong Provincial People's Hospital. The study evaluate the efficacy of oral magnesium L-threonate supplementation on improving menopausal symptoms and quality of life among peri/post-menopausal women.

This trial aims to explore whether oral magnesium L-threonate supplementation could alleviate menopausal syndromes.

Participants will randomly assigned to conduct oral magnesium L-threonate supplementation or placebo for 8 weeks. Face-to-face and internet follow up will be conducted once per 2 weeks.

DETAILED DESCRIPTION:
The peri-menopausal period is a crucial transitional stage for women from middle age to old age. During this period, there is a dramatic and continuous decline in estrogen levels in women's bodies. The rapid change in estrogen levels triggers a series of complex physiological and pathological changes, leading to many clinical symptoms in perimenopausal women. The menopausal syndrome encompasses osteoporosis and joint-muscle pain, hot flashes and night sweats in terms of vasomotor symptoms, mood swings and memory loss, etc. It greatly troubles women physically and mentally and affects their daily lives. Currently, the main treatment methods for menopausal syndrome include hormone replacement therapy (HRT) and selective serotonin reuptake inhibitors (SSRI). However, both of these treatment methods are accompanied by significant side effects. Hormone replacement therapy may increase the risk of diseases such as breast cancer, endometrial cancer, and venous thrombosis. Therefore, there is an urgent need to explore safe and effective new therapies to improve the health of perimenopausal women.

Magnesium ions, as important cations in the human body, play an indispensable role in maintaining the normal physiological functions of the body. In perimenopausal women, due to the decrease in estrogen levels, the level of magnesium is greatly decreased. Magnesium deficiency not only aggravates the symptoms of menopausal syndrome but also may increase the risk of chronic diseases such as cardiovascular diseases and osteoporosis.

However, traditional magnesium supplements, such as magnesium sulfate and magnesium oxide, have obvious limitations in practical applications. After oral administration, traditional magnesium supplements cannot effectively increase the intracellular magnesium concentration, and cannot cross the blood-brain barrier and are difficult to act on the nervous system to improve pain, hot flashes, and other menopausal symptoms.

Magnesium L - threonate is a new magnesium supplement with unique advantages. It is an oral preparation that can effectively supplement intracellular magnesium. Its greatest feature is that it can smoothly cross the blood-brain barrier and directly act on the central nervous system. Although it has been proven to be relatively safe, currently, the randomized controlled trials related to magnesium L - threonate have only confirmed its improvement effects on pain and cognitive function [23,24], and the research on its effect on improving overall menopausal symptoms is rare.

This study aims to deeply explore whether magnesium L-threonate can effectively improve the menopausal symptoms of perimenopausal women and improve their quality of life.

Participants will be randomly divided into an intervention group and a control group, and medications are administered according to the following protocols:

Intervention group: Magnesium L-threonate, 1740 mg, taken orally, twice a day, for 8 weeks.

Control group: Placebo of magnesium L-threonate, 1740 mg, taken orally, twice a day, for 8 weeks.

The face-to-face questionnaire surveys, physical examinations, and biological sample collections will be conducted during the study screening period and at the end of the study (8 weeks completed) ± 1 day. The online questionnaire surveys will be carried out on the 3rd week ± 1 day, 5th week ± 1 day, and 7th week ± 1 day of the intervention period.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 40-60 years;
2. Postmenopausal status or in the late menopausal transition stage. 3. Postmenopausal status is defined as: natural menopause with no menstruation in the past 12 months. The late menopausal transition stage will be defined as: amenorrhea for at least 60 days within the past 12 months;

4. MRS score ≥15 points based on symptoms in the past 1 month; 5. Willing to complete the required follow-up visits during the trial period. 6. Voluntarily sign the informed consent form.

Exclusion Criteria:

1. History of bilateral oophorectomy or hysterectomy;
2. Current or past use of magnesium L-threonate preparations or similar nutrient formulations within the last 3 months;
3. Definite history of gastrointestinal diseases that may affect the absorption of the investigational drug;
4. Definite history of liver diseases that may affect the metabolism of the investigational drug;
5. Definite history of kidney diseases that may affect the excretion of the investigational drug, with serum creatinine levels > 2 mg/dL (88.4 μmol/L);
6. Current or recent use of hormone replacement therapy: vaginal or transdermal estrogen within the past 4 weeks; oral estrogen or progesterone within the past 8 weeks; intrauterine progesterone therapy within the past 8 weeks; progesterone implants or estrogen injection therapy within the past 3 months; estrogen pellet therapy or progesterone injection therapy within the past 6 months; or intention to use these medications during the intervention period;
7. Current or past use of medications such as clonidine, methyldopa, gabapentin, pregabalin, and selective serotonin or norepinephrine reuptake inhibitors (SSRIs/SNRIs) within the past 1 month, or intention to use these medications during the intervention period;
8. Current or past use of phosphodiesterase inhibitor medications within the past 1 month, or intention to use these medications during the intervention period;
9. Autoimmune diseases requiring medication, current or past treatment with glucocorticoids, antirheumatic drugs, or biologics within the past 6 months, or intention to use these medications during the intervention period;
10. Depression or anxiety requiring medication, current or past use of antidepressants within the past 3 months, or intention to use these medications or treatments during the intervention period;
11. Current or past use of hypnotic medications such as diazepam or triazolam within the past 2 weeks, or intention to use these medications during the intervention period;
12. Osteoarthritis, osteoporosis, or other musculoskeletal diseases requiring medication;
13. Known allergy to magnesium L-threonate;
14. History of malignancy, or life expectancy less than 1 year;
15. Major surgery within the past 6 months, or intention to undergo surgery during the intervention period, including but not limited to cardiac surgery or joint replacement;
16. Currently pregnant, having given birth within the past 3 months, planning pregnancy during the study period, or unwilling to use conventional barrier contraception or abstain from sexual activity to prevent pregnancy if not fully menopausal;
17. Currently breastfeeding, having breastfed within the past 3 months, or planning to breastfeed during the study period;
18. Unable or unwilling to provide informed consent, complete questionnaires, or attend study visits;
19. Participation in other interventional studies;
20. Other conditions judged by the investigator as unsuitable for trial participation. These conditions may make potential participants highly unlikely to adhere to the study protocol, including plans to relocate, substance abuse, severe psychiatric issues, or severe dementia.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of Menopausal Rating Scale (MRS) | From randomization to the end of treatment at 8 weeks
  The Menopausal Rating Scale (MRS) is a widely used tool for assessing the severity of menopausal symptoms and their impact on a woman's quality of life (Health Qual Life Outcomes 2004;2:67). The MRS consists of multiple domains and specific items. Typically, it includes categories such as somatic symptoms (like hot flashes, sweating, sleep disturbances), psychological symptoms (including mood swings, anxiety, and depression), and urogenital symptoms (such as vaginal dryness and urinary problems). Each item within these domains is scored on a numerical scale, usually ranging from 0 to 3 or 0 to 4, depending on the severity of the symptom, and the maximum total score would be 44. A score of 0 often indicates the absence of the symptom, while higher scores reflect increasing levels of discomfort or impairment.

SECONDARY OUTCOMES:
Change of Menopause Quality of Life (MENQOL) Questionnaire | From randomization to the end of treatment at 8 weeks
  The Menopause Quality of Life Questionnaire (MENQOL) assesses the impact of menopausal symptoms across four domains: vasomotor, sexual, physical, and psychosocial (Maturitas 24:161-175, 1996). Symptoms like hot flashes, vaginal dryness, and depression are evaluated. Participants first indicate if they've had symptoms in the past month, then rate bothersomeness on a 7-point scale. Ratings are recorded from 2 (symptom present but not bothersome) to 8 (extremely bothered). Domain scores are calculated as the mean of item scores; higher scores mean more troublesome symptoms and poorer quality of life. The score of MENQOL Questionnaire is from 8 to 232.
Change of EuroQoL 5-dimension 5-Level (EQ5D-5L) | From randomization to the end of treatment at 8 weeks
  The EQ-5D 5-Level (EuroQol Five Dimensions) is a standardized questionnaire designed to measure health status and health-related quality of life (Qual Life Res 2011;20:1727-36). It evaluates five dimensions: mobility, self-care, usual activities (e.g., work, housework), pain/discomfort, and anxiety/depression. Scoring Ranges
  EQ-VAS (Visual Analog Scale):
  Range: 0-100. Interpretation: 0 represents the worst imaginable health state, and 100 represents the best possible health state. This scale reflects the respondent's self-assessment of overall health.
  EQ-5D Index Score (Utility Value):
  Range: 0 to 1.
  Interpretation:
  1: Perfect health. 0: Equivalent to death. Negative values: Worse than death (e.g., severe chronic conditions).
Change of Brief Pain Inventory-Short Form (BPI-SF) | From randomization to the end of treatment at 8 weeks
  The Brief Pain Inventory-Short Form (BPI-SF) is a widely used tool for assessing pain (Pain. 1983;17(2): 197-210). This 14-item questionnaire requires respondents to rate their joint pain experienced over the past week and the extent to which the pain disrupts their activities. Ratings are given on a scale of 0 to 10, where 0 indicates "no pain" and 10 represents "pain as severe as imaginable". The range of the score number is from 0 to 140 points.
Change of Hot flash Score | From randomization to the end of treatment at 8 weeks
  The Hot Flash Score was measured using a prospective, self-report hot flash diary, which women were instructed to fill out in real-time (J Clin Oncol 19:4280-4290, 2001). The determination of hot flash scores involved allocating points to each hot flash according to the reported severity. Specifically, a hot flash was assigned 1 point for mild severity, 2 points for moderate severity, 3 points for severe severity, and 4 points for very severe severity. For each patient, the points assigned to hot flashes on each day were summed up, and then these daily totals were averaged over each week of the trial period. The minimum of the score is 0, and there is no maximum limit.
Change of Insomnia Severity Index（ISI） | From randomization to the end of treatment at 8 weeks
  The Insomnia Severity Index (ISI) is a self-rated questionnaire designed to assess the severity of insomnia (Sleep Med. 2001;2:297-307). It is used to evaluate various aspects of insomnia, including difficulty falling asleep, staying asleep, early morning awakening, and the impact of insomnia on daytime functioning and well - being.
  The ISI consists of 7 items, and each item is scored on a scale of 0-4. So the total score of the ISI ranges from 0 to 28.
  A score of 0-7 indicates no clinically significant insomnia. A score of 8-14 suggests sub - threshold insomnia. A score of 15-21 represents moderate insomnia. A score of 22-28 indicates severe insomnia.
Change of Self-Rating Depression Scale（SDS） | From randomization to the end of treatment at 8 weeks
  The Self-Rating Depression Scale (SDS) is a self-administered psychological assessment tool used to measure the severity of depressive symptoms in individuals (Arch Gen Psychiatry. 1973;29(3):328-337). The scale contains 20 statements related to common symptoms of depression, such as mood, sleep, appetite, and self-esteem. Respondents rate each statement according to how often they have experienced the described symptom in the past week, using a 4-point scale: 1 (rarely), 2 (sometimes), 3 (mostly), and 4 (almost always).The total raw score of the SDS ranges from 20 (the lowest possible score, indicating no depressive symptoms) to 80 (the highest possible score, suggesting severe depressive symptoms).
Change of Generalized Anxiety Disorder 7-item scale (GAD-7) | From randomization to the end of treatment at 8 weeks
  The Generalized Anxiety Disorder 7 - item scale (GAD-7) is a brief self-report questionnaire designed to screen for generalized anxiety disorder and assess the severity of anxiety symptoms (Archives of Internal Medicine, 166(10), 1092-1097). It consists of 7 items related to common symptoms of anxiety, such as feeling nervous, worried, or on edge; not being able to stop or control worrying; and having trouble relaxing.
  Each item is scored on a 4 - point scale: 0 (Not at all), 1 (Several days), 2 (More than half the days), and 3 (Nearly every day). The total score of the GAD-7 ranges from 0 to 21.
  A score of 0-4 is generally considered to indicate minimal anxiety. A score of 5-9 suggests mild anxiety. A score of 10-14 indicates moderate anxiety. A score of 15-21 represents severe anxiety.
Change of IL-6 level | From randomization to the end of treatment at 8 weeks
Change of hsCRP level | From randomization to the end of treatment at 8 weeks
Change of P1NP level | From randomization to the end of treatment at 8 weeks
Change of N-CTX level | From randomization to the end of treatment at 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Global Health Research Center,Guangdong Provincial People's Hospital(Guanadong Academy of Medical Sciences), Guangzhou, Guangdong, China